CLINICAL TRIAL: NCT06340529
Title: Comparison of the Perception of Non-technical Skills by Students, Self-assessment and Teachers, Developed During the Clinical Simulation in Students of the Degree in Physiotherapy
Brief Title: Comparison of the Perception of Non-technical Skills
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, María del Carmen Casal Angulo, Principal investigator, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CLS_SIMULATION
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Physioterapy; Students; Clinical Simulation; Learning methodology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Between equals (Active Comparator): Physiotherapy students who do not participate in the simulation, but they do observe the simulation and participate in the debriefing.
  Interventions: Other: Clinical Simulation
- Self appraisal (Experimental): Physiotherapy students who participate in the simulation in all its phases.
  Interventions: Other: Clinical Simulation
- Lecturers (Active Comparator): Teachers observing the intervention and participate as patients and in the debriefing
  Interventions: Other: Clinical Simulation

INTERVENTIONS:
Other: Clinical Simulation — Carrying out a total of 9 clinical simulation in three days, one day every two weeks, where the student resolves a situation by taking on the role of a physiotherapist with a simulated patient.

SUMMARY:
Clinical simulation has recently acquired great importance in the health sciences. It is a pedagogical methodology that is increasingly used in health science degrees, since it is very useful for the acquisition of both technical and non-technical skills (leadership, teamwork and effective communication, among others).

However, if the investigators focus on physical therapy, the use of clinical simulation is a novel field and therefore requires a great deal of research. Researchers in this field do not yet have the consistency and experience as in other health branches such as medicine or nursing, where the participants have been using high-fidelity simulators for years for the learning of all their students.

Clinical simulation allows students to achieve these competencies without the need to practice on real patients. For all these reasons, and because of the situation of need generated in recent years, in which internships in hospitals and clinical centers were completely suppressed, the need for our research is justified.

ELIGIBILITY:
Inclusion Criteria:

* Second year students of the Physiotherapy Degree
* They do not have clinical experience with real patients.
* Subject teachers

Exclusion Criteria:

* Not wanting to sign to participate in the study.
* Not signing the informed consent
* Teachers who do not have experience in clinical simulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Ottawa Scale | 2 week, 4 week, 6 week.
  Modified Ottawa Scale for the acquisition of non-technical skills, validated in Spanish (https://doi.org/10.1016/j.redar.2021.02.009).
  Each of the items evaluated must is be classified from 'strongly disagree', whose value is one, to 'strongly agree', whose value is 7. The minimum value is six and maximum value is forty-two. Higher scores mean a better outcome.
  The scale will be passed after each of the 9 simulations.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Casal-Angulo, PhD RN, Study Director — University of Valencia
Locations (1):
- Carmen Casal, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No